CLINICAL TRIAL: NCT01581541
Title: Phase I Study of the Hsp90 Inhibitor, PU-H71, in Patients With Refractory Solid Tumors and Low-Grade Non-Hodgkin's Lymphoma
Brief Title: PU-H71 in Patients With Solid Tumors and Low-Grade Non-Hodgkin's Lymphoma That Have Not Responded to Standard Treatment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study closed prematurely due to discontinuation of drug supply.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alice Chen, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 110150; 11-C-0150
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Solid Tumors; Lymphoma
Keywords: Targeted Therapy; Solid Tumors; Lymphoma; Non-Hodgkin Lymphoma; Solid Tumor
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — 9H-purine-9-propanamine, 6-amino-8-((6-iodo-1,3-benzodioxol-5-yl)thio)-N-(1-methylethyl)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PU-H71 (Experimental): PU-H71 will be administered intravenous (IV) over one hour, once weekly, 2 weeks out of 3, (i.e., on days 1 and 8) every 21 days
  Interventions: Drug: PU-H71

INTERVENTIONS:
Drug: PU-H71 — PU-H71 is a synthetic HSP90 inhibitor which can bind both open and closed conformations of HSP90. It demonstrates extended tumor retention and client protein degradation, while being rapidly cleared from normal tissues. It has shown complete tumor responses and retained sensitivity to retreatment in vivo.

SUMMARY:
Background:

- PU-H71 is an experimental drug used to treat cancer. It works by blocking a protein in tumors. When this protein is blocked, it affects other proteins inside the cell that cancers need to grow. Researchers want to study whether PU-H71 is a safe and effective way to treat solid tumors and non-Hodgkin's lymphoma.

Objectives:

- To evaluate the safety and effectiveness of PU-H71 in solid tumors and non-Hodgkin's lymphoma that have not responded to standard treatments.

Eligibility:

- Individuals at least 18 years of age who have solid tumors or non-Hodgkin's lymphoma that have not responded to standard treatments.

Design:

* Patients will be screened with a physical exam, medical history, blood tests, and imaging studies.
* Patients will receive PU-H71 as a 1-hour dose on days 1 and 8 of a 21-day cycle of treatment. The first treatment cycle will be done in the hospital so that patients can be monitored. The next treatment cycles will be done on an outpatient basis.
* Patients will have blood and urine tests and eye exams.
* Patients will provide tumor samples for study.
* Patients will have imaging studies to monitor tumor response to treatment.
* Patients will continue to take PU-H71 for as long as side effects remain tolerable and their tumor or lymphoma does not worsen. Study researchers may adjust the dose if needed.

DETAILED DESCRIPTION:
Background:

-PU-H71 is a synthetic HSP90 inhibitor which can bind both open and closed conformations of HSP90. It demonstrates extended tumor retention and client protein degradation, while being rapidly cleared from normal tissues. It has shown complete tumor responses and retained sensitivity to retreatment in vivo.

Primary Objectives:

* To establish the safety and tolerability of PU-H71 administered on a once weekly, 2 weeks out of 3 schedule, in patients with refractory solid tumors and lowgrade non-Hodgkin's lymphoma (NHL).
* To establish the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of PU-H71 administered on a once weekly, 2 weeks out of 3 schedule, in patients with refractory solid tumors and low-grade NHL.
* To determine the pharmacokinetics of PU-H71 administered on a once weekly, 2 weeks out of 3 schedule, in patients with refractory solid tumors and low-grade NHL.

Secondary Objectives:

* To perform pharmacodynamic studies to ascertain PU-H71 effect on HSP70 in tumor tissue, serum, and peripheral blood mononuclear cells (PBMCs) at the MTD.
* To perform pharmacodynamic studies to ascertain PU-H71 effect on HSP90 client proteins in tumor tissue at the MTD.

Eligibility:

-Study participants must have histologically confirmed solid tumor malignancy or low-grade non-Hodgkin s lymphoma that has progressed or recurred after at least one line of chemotherapy or for which no standard treatment option exists; no therapy within 4 weeks prior to entering the study; age greater than or equal to 18 years; Eastern Cooperative Oncology Group (ECOG) less than or equal to 2; life expectancy > 3 months; and adequate organ and marrow function. Patients entering on the expansion cohort at the MTD must have disease amenable to biopsy with willingness to undergo pre- and post-treatment biopsies.

Study Design:

* This study will follow a modified accelerated titration design (Simon et al., 1997).
* The accelerated phase ends when 1 patient experiences a dose-limiting toxicity or 2 patients experience Grade 2 drug-related toxicity during the first cycle; after which the study will follow the standard 3 + 3 design.
* PU-H71 will be administered intravenously over one hour, once weekly, 2 weeks out of 3, (i.e., on days 1 and 8) every 21 days.
* Pharmacokinetics (PK) and pharmacodynamics (PD) studies will be conducted during cycle 1. Up to 10 additional patients will be entered at the MTD to further define toxicity and perform PD studies at this dose; pre- and post-treatment tumor biopsies will be mandatory for these patients.
* Computed tomography (CT) scans will be performed at baseline and every 2 cycles (6 weeks) for restaging.
* Up to 100 patients may be treated.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically documented (confirmed at the Laboratory of Pathology, National Cancer Institute (NCI)) solid tumor malignancy or low-grade non-Hodgkin's lymphoma that is metastatic or unresectable, for which standard curative measures do not exist, or whose disease has progressed or recurred following at least one line of standard therapy.
* Patients must have measurable or evaluable disease.
* Patients must have completed any chemotherapy, radiation therapy, or biologic therapy greater than or equal to 4 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin C).

Patients must be greater than or equal to 2 weeks since any prior administration of a study drug in a Phase 0 study (also referred to as a pre-Phase I study where a sub-therapeutic dose of drug is administered). Patients must have recovered to eligibility levels from prior toxicity or adverse events. Patients receiving bisphosphonates for any cancer are eligible to participate.

* Age greater than or equal to 18 years.
* An Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Life expectancy > 3 months.
* Patients must have normal or adequate organ and marrow function as defined below:

  * Absolute neutrophil count greater than or equal to 1,500/microL
  * Platelets greater than or equal to 100,000/microL
  * Total bilirubin less than or equal to 1.5 times institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST)serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic pyruvic transaminase(SGPT) less than or equal to 2.5 times institutional ULN
  * Creatinine <1.5 times ULN; OR
  * Measured creatinine greater than or equal to 60 mL/minute for patients with clearance creatinine levels greater than or equal to 1.5 times ULN
* The effects of PU-H71 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry, for the duration of study participation, and for 2 months after completion of study. Women of childbearing potential must have a negative pregnancy test within 72 hours of enrollment in order to be eligible. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in the study, the treating physician should be notified immediately. Because there is an unknown but potential risk to nursing infants secondary to treatment of the mother with PU-H71, breastfeeding should be discontinued if the mother is treated with PU-H71.
* During the expansion phase of the protocol, patients must have:

  * Disease amenable to biopsy
  * Willingness to undergo pre- and post-treatment tumor biopsies
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients with known brain metastases or carcinomatous meningitis are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status has remained stable for greater than or equal to 3 months after treatment of the brain metastases.
* Patients with clinically significant intercurrent illnesses, including but not limited to, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Corrected QT interval (QTc) > 450 msec for men and > 470 msec for women.
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetics (PK) interactions with PU-H71.
* Pregnant women are ineligible because the effects of PU-H71 on the developing human fetus are unknown. Breastfeeding should be discontinued if the mother is treated with PU-H71 since there is an unknown but potential risk for adverse events in nursing infants.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-04-26 (Actual); Primary Completion 2014-09-03 (Actual); Study Completion 2014-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zuehlke A, Johnson JL. Hsp90 and co-chaperones twist the functions of diverse client proteins. Biopolymers. 2010 Mar;93(3):211-7. doi: 10.1002/bip.21292. PMID 19697319
- [Background] Fukuyo Y, Hunt CR, Horikoshi N. Geldanamycin and its anti-cancer activities. Cancer Lett. 2010 Apr 1;290(1):24-35. doi: 10.1016/j.canlet.2009.07.010. Epub 2009 Oct 21. PMID 19850405
- [Background] Chavany C, Mimnaugh E, Miller P, Bitton R, Nguyen P, Trepel J, Whitesell L, Schnur R, Moyer J, Neckers L. p185erbB2 binds to GRP94 in vivo. Dissociation of the p185erbB2/GRP94 heterocomplex by benzoquinone ansamycins precedes depletion of p185erbB2. J Biol Chem. 1996 Mar 1;271(9):4974-7. doi: 10.1074/jbc.271.9.4974. PMID 8617772
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0150.html

RESULTS

PARTICIPANT FLOW:
Groups:
- PU-H71, 10 mg/m^2: PU-H71 will be administered intravenous (IV) over one hour, once weekly, 2 weeks out of 3, (i.e., on days 1 and 8) every 21 days
- PU-H71, 20 mg/m^2; PU-H71, 40 mg/m^2; PU-H71, 60 mg/m^2; PU-H71, 80 mg/m^2; PU-H71, 110 mg/m^2; PU-H71, 150 mg/m^2; PU-H71, 200 mg/m^2; PU-H71, 266 mg/m^2; PU-H71, 354 mg/m^2; PU-H71, 470 mg/m^2: PU-H71 will be administered IV over one hour, once weekly, 2 weeks out of 3, (i.e., on days 1 and 8) every 21 days
Period: Overall Study
Arm/Group | PU-H71, 10 mg/m^2 | PU-H71, 20 mg/m^2 | PU-H71, 40 mg/m^2 | PU-H71, 60 mg/m^2 | PU-H71, 80 mg/m^2 | PU-H71, 110 mg/m^2 | PU-H71, 150 mg/m^2 | PU-H71, 200 mg/m^2 | PU-H71, 266 mg/m^2 | PU-H71, 354 mg/m^2 | PU-H71, 470 mg/m^2
Started | 1 | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 1 | 3 | 1
Completed | 1 | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 1 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | PU-H71
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 59 [19 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17
Number of Prior Therapies [Mean (Full Range); unit: prior therapies] | 7 [1 to 14]
Diagnosis [Count of Participants; unit: Participants]
  Malignant Hürthle cell tumor | 1
  Rectal adenocarcinoma | 1
  Adenocarcinoma, not otherwise specified | 6
  Adenoid cystic carcinoma | 1
  Invasive poorly differentiated carcinoma | 1
  Metastatic adenocarcinoma | 1
  Hepatocellular carcinoma | 1
  Carcinoid tumor | 1
  Squamous cell carcinoma of the esophagus | 1
  Synovial sarcoma | 2
  Non-small cell lung cancer | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cycle 1 Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as an adverse event that occurred during cycle 1, was thought to be related to study drug administration, and met one of the following criteria: grade ≥ 3 non-hematologic toxicities (except diarrhea, nausea, vomiting without maximal supportive therapy; alopecia), grade 4 hematologic toxicities (except lymphopenia), and grade 2 ocular toxicity that did not resolve to ≤ grade 1 within 2 weeks. Occurrence of a DLT resulted in a dose reduction following resolution to grade ≤ 2. No more than 2 dose reductions were allowed per patient on study.
Time Frame: Cycle 1 (21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | PU-H71, 10 mg/m^2 | PU-H71, 20 mg/m^2 | PU-H71, 40 mg/m^2 | PU-H71, 60 mg/m^2 | PU-H71, 80 mg/m^2 | PU-H71, 110 mg/m^2 | PU-H71, 150 mg/m^2 | PU-H71, 200 mg/m^2 | PU-H71, 266 mg/m^2 | PU-H71, 354 mg/m^2 | PU-H71, 470 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 1 | 3 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events Possibly, Probably, or Definitely Related to Study Drug
Description: Severity of adverse events were graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Grade 1 Mild adverse event (AE), Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, and Grade 5 Death related to AE.
Time Frame: 3 years and two months and 11 days
Measure: Count of Participants; unit: Participants
Arm/Group | PU-H71, 10 mg/m^2 | PU-H71, 20 mg/m^2 | PU-H71, 40 mg/m^2 | PU-H71, 60 mg/m^2 | PU-H71, 80 mg/m^2 | PU-H71, 110 mg/m^2 | PU-H71, 150 mg/m^2 | PU-H71, 200 mg/m^2 | PU-H71, 266 mg/m^2 | PU-H71, 354 mg/m^2 | PU-H71, 470 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 1 | 3 | 1
Participants
  Grade 2 Anemia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Grade 2 Aspartate Aminotransferase | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 Atrioventricular Block First Degree | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Blood Bilirubin Increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 Fatigue | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Headache | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Lymphopenia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 Nausea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Sinus Bradycardia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Vomiting | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Maximum Tolerated Dose (MTD) of PU-H71
Description: The MTD is the dose level at which no more than 1 of 6 patients experience DLT during the first cycle of treatment, and the dose below that at which at least 2 (of ≤ 6) patients have DLT as a result of the drug.
Time Frame: Cycle 1 (21 days)
Measure: Number; unit: mg/m^2
Arm/Group | PU-H71
Number analyzed (Participants) | 17
mg/m^2 | NA — Due to cessation of the drug supply, patients could not be accrued at higher doses, and the MTD could not be determined.

4. Secondary Outcome: Number of Participants According to Best Response Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1)
Description: Number of Participants According to Best Response Per Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by computed tomography (CT): Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (POD); POD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions.
Time Frame: Baseline and every 6 weeks up to 18 weeks
Population: All participants who continued further treatment and did not start an alternative treatment were considered evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | PU-H71, 10 mg/m^2 | PU-H71, 20 mg/m^2 | PU-H71, 40 mg/m^2 | PU-H71, 60 mg/m^2 | PU-H71, 80 mg/m^2 | PU-H71, 110 mg/m^2 | PU-H71, 150 mg/m^2 | PU-H71, 200 mg/m^2 | PU-H71, 266 mg/m^2 | PU-H71, 354 mg/m^2 | PU-H71, 470 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 3 | 1 | 1 | 1 | 2 | 1
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 0
  Progression of Disease | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1

5. Secondary Outcome: Number of Days on Treatment
Time Frame: up to 126 days
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | PU-H71, 10 mg/m^2 | PU-H71, 20 mg/m^2 | PU-H71, 40 mg/m^2 | PU-H71, 60 mg/m^2 | PU-H71, 80 mg/m^2 | PU-H71, 110 mg/m^2 | PU-H71, 150 mg/m^2 | PU-H71, 200 mg/m^2 | PU-H71, 266 mg/m^2 | PU-H71, 354 mg/m^2 | PU-H71, 470 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 3 | 1 | 1 | 1 | 2 | 1
days | 42 [42 to 42] | 42 [42 to 42] | 42 [42 to 42] | 84 [84 to 84] | 42 [42 to 42] | 126 [42 to 126] | 84 [84 to 84] | 84 [84 to 84] | 63 [63 to 63] | 42 [42 to 42] | 42 [42 to 42]

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The maximum concentration (Cmax) was determined by visual inspection of the concentration versus time data.
Time Frame: Before the start of infusion, 30 minutes after the start of infusion, 5 minutes before completion of infusion, and at 1.5, 2, 3, 4, 7, 10, and 24 hours after the start of infusion on day 1 during cycle 1.
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | PU-H71, 10 mg/m^2 | PU-H71, 20 mg/m^2 | PU-H71, 40 mg/m^2 | PU-H71, 60 mg/m^2 | PU-H71, 80 mg/m^2 | PU-H71, 110 mg/m^2 | PU-H71, 150 mg/m^2 | PU-H71, 200 mg/m^2 | PU-H71, 266 mg/m^2 | PU-H71, 354 mg/m^2 | PU-H71, 470 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 1 | 3 | 1
µM | 0.2 (0) | 0.3 (0) | 74.7 (0) | 1.3 (0) | 5.17 (0.1) | 7.3 (2.4) | 8.7 (0) | 8.0 (4.5) | 7.8 (0) | 17.3 (8.5) | 33.7 (0)

7. Secondary Outcome: Terminal Half-life (T1/2)
Description: The terminal half-life (t1/2) was derived from the plasma concentration vs. time data.
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PU-H71, 10 mg/m^2 | PU-H71, 20 mg/m^2 | PU-H71, 40 mg/m^2 | PU-H71, 60 mg/m^2 | PU-H71, 80 mg/m^2 | PU-H71, 110 mg/m^2 | PU-H71, 150 mg/m^2 | PU-H71, 200 mg/m^2 | PU-H71, 266 mg/m^2 | PU-H71, 354 mg/m^2 | PU-H71, 470 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 1 | 3 | 1
hours | 2.7 (0) | 10.5 (0) | 9.2 (0) | 6.1 (0) | 6.7 (0.1) | 7.6 (0.2) | 7.2 (0) | 7.1 (0.5) | 10.2 (0) | 11.5 (7.3) | 10.8 (0)

8. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to 24 Hours [AUC(0-24)]
Description: Area Under the Concentration-Time Curve From Time 0 to 24 Hours was estimated by trapezoidal rule calculations
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: µM*min
Arm/Group | PU-H71, 10 mg/m^2 | PU-H71, 20 mg/m^2 | PU-H71, 40 mg/m^2 | PU-H71, 60 mg/m^2 | PU-H71, 80 mg/m^2 | PU-H71, 110 mg/m^2 | PU-H71, 150 mg/m^2 | PU-H71, 200 mg/m^2 | PU-H71, 266 mg/m^2 | PU-H71, 354 mg/m^2 | PU-H71, 470 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 1 | 3 | 1
µM*min | 27 (0) | 74 (0) | 3845 (0) | 273 (0) | 899 (32) | 1186 (481) | 1534 (0) | 2090 (459) | 3596 (0) | 6866 (2876) | 8568 (0)

9. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity [AUC(0-∞)]
Description: Area Under the Concentration-Time Curve From Time 0 to Infinity was estimated by trapezoidal rule calculations
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: µM*min
Arm/Group | PU-H71, 10 mg/m^2 | PU-H71, 20 mg/m^2 | PU-H71, 40 mg/m^2 | PU-H71, 60 mg/m^2 | PU-H71, 80 mg/m^2 | PU-H71, 110 mg/m^2 | PU-H71, 150 mg/m^2 | PU-H71, 200 mg/m^2 | PU-H71, 266 mg/m^2 | PU-H71, 354 mg/m^2 | PU-H71, 470 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 1 | 3 | 1
µM*min | 31 (0) | 100 (0) | 3905 (0) | 301 (0) | 1007 (32) | 1375 (591) | 1771 (0) | 2477 (429) | 5449 (0) | 10815 (5499) | 12151 (0)

10. Secondary Outcome: Urinary Excretion (%)
Description: Elimination of the drug was investigated by analysis of an aliquot of the total urine collected in 24 h.
Time Frame: Every void post-treatment on day 1 of cycle 1
Measure: Mean (Standard Deviation); unit: percent of dose recovered
Arm/Group | PU-H71, 10 mg/m^2 | PU-H71, 20 mg/m^2 | PU-H71, 40 mg/m^2 | PU-H71, 60 mg/m^2 | PU-H71, 80 mg/m^2 | PU-H71, 110 mg/m^2 | PU-H71, 150 mg/m^2 | PU-H71, 200 mg/m^2 | PU-H71, 266 mg/m^2 | PU-H71, 354 mg/m^2 | PU-H71, 470 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 1 | 3 | 1
percent of dose recovered | 5.5 (0) | NA (NA) — Data were not collected from the single participant at this dose level. | 1.9 (0) | 8.8 (0) | 6.7 (1.3) | 6.7 (4.6) | 8.1 (0) | 6.0 (4.2) | 5.4 (0) | 8.6 (4.6) | 5.7 (0)

11. Secondary Outcome: Clearance
Description: Clearance was calculated from drug dose and AUC(0-∞).
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/h/kg
Arm/Group | PU-H71, 10 mg/m^2 | PU-H71, 20 mg/m^2 | PU-H71, 40 mg/m^2 | PU-H71, 60 mg/m^2 | PU-H71, 80 mg/m^2 | PU-H71, 110 mg/m^2 | PU-H71, 150 mg/m^2 | PU-H71, 200 mg/m^2 | PU-H71, 266 mg/m^2 | PU-H71, 354 mg/m^2 | PU-H71, 470 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 1 | 3 | 1
L/h/kg | 1.03 (0) | 0.63 (0) | 0.03 (0) | 0.63 (0) | 0.25 (0.01) | 0.28 (0.12) | 0.27 (0) | 0.26 (0.04) | 0.15 (0) | 0.13 (0.09) | 0.12 (0)

ADVERSE EVENTS:
Time Frame: 3 years and two months and 11 days
Description: Adverse events were collected and analyzed by dose level.
Arm/Group | PU-H71, 10 mg/m^2 | PU-H71, 20 mg/m^2 | PU-H71, 40 mg/m^2 | PU-H71, 60 mg/m^2 | PU-H71, 80 mg/m^2 | PU-H71, 110 mg/m^2 | PU-H71, 150 mg/m^2 | PU-H71, 200 mg/m^2 | PU-H71, 266 mg/m^2 | PU-H71, 354 mg/m^2 | PU-H71, 470 mg/m^2
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 1/1 | 1/1 | 0/2 | 0/3 | 0/1 | 0/2 | 1/1 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 0/1 | 0/1 | 0/2 | 0/3 | 0/1 | 0/2 | 0/1 | 1/3 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 2/2 | 3/3 | 1/1 | 2/2 | 1/1 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PU-H71, 10 mg/m^2 (N=1) | PU-H71, 20 mg/m^2 (N=1) | PU-H71, 40 mg/m^2 (N=1) | PU-H71, 60 mg/m^2 (N=1) | PU-H71, 80 mg/m^2 (N=2) | PU-H71, 110 mg/m^2 (N=3) | PU-H71, 150 mg/m^2 (N=1) | PU-H71, 200 mg/m^2 (N=2) | PU-H71, 266 mg/m^2 (N=1) | PU-H71, 354 mg/m^2 (N=3) | PU-H71, 470 mg/m^2 (N=1)
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PU-H71, 10 mg/m^2 (N=1) | PU-H71, 20 mg/m^2 (N=1) | PU-H71, 40 mg/m^2 (N=1) | PU-H71, 60 mg/m^2 (N=1) | PU-H71, 80 mg/m^2 (N=2) | PU-H71, 110 mg/m^2 (N=3) | PU-H71, 150 mg/m^2 (N=1) | PU-H71, 200 mg/m^2 (N=2) | PU-H71, 266 mg/m^2 (N=1) | PU-H71, 354 mg/m^2 (N=3) | PU-H71, 470 mg/m^2 (N=1)
Abdominal pain - cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 | 1 (2) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain - Left (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (2) | 1 (3) | 1 (7) | 2 (3) | 3 (8) | 1 (4) | 2 (2) | 0 (0) | 3 (4) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection, device related (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 2 (3) | 1 (3)
Night blindness: intermittent (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity- Right Ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral vascular dis. (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No